CLINICAL TRIAL: NCT05858372
Title: Effects of Chios Mastiha Essential Oil on Cholesterol Levels of Healthy Volunteers: a Prospective, Randomized, Placebo-controlled Study (MASTIHA-OIL Study)
Brief Title: Effects of Chios Mastiha Essential Oil on Cholesterol Levels of Healthy Volunteers
Acronym: MASTIHA-OIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHEPA University Hospital (Other)
Collaborators: Skylitseio General Hospital of Chios (Unknown)
Responsible Party: Principal Investigator, Matthaios Didagelos, Cardiologist, AHEPA University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-19/02/2020
Record Dates: First submitted 2023-05-04; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Hyperlipidemias; Hypercholesterolemia
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chios Mastiha essential oil (Experimental): 1 soft gel capsule containing 200 mg of CMO and 100 mg of other excipients being medium chain triglycerides, while the shell was made of bovine gelatin and glycerol
  Interventions: Dietary Supplement: Chios Mastiha essential oil
- Placebo (Placebo Comparator): 1 soft gel capsule only 100 mg of other excipients being medium chain triglycerides, while the shell was made of bovine gelatin and glycerol
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Chios Mastiha essential oil — 1 soft gel capsule containing 200 mg of CMO and 100 mg of other excipients being medium chain triglycerides, while the shell was made of bovine gelatin and glycerol
  Arms: Chios Mastiha essential oil
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A prospective, randomized, placebo-controlled study was designed to study the hypolipidemic effect of CMO capsules on healthy volunteers with elevated cholesterol levels.

DETAILED DESCRIPTION:
Background Chios Mastiha essential oil (CMO) is a natural product extracted from the resin of Mastiha, possessing antioxidant, anti-microbial, anti-ulcer,anti-neoplasmatic and cholesterol lowering capabilities in vitro, and its hypolipidemic effect was confirmed in animal studies. Yet, there are no randomized, placebo-controlled clinical studies in the literature regarding CMO's hypolipidemic effects in humans.

Design A prospective, randomized, placebo-controlled study was designed to study the hypolipidemic effect of CMO capsules on healthy volunteers with elevated cholesterol levels.

Methods 192 healthy volunteers were screened and eventually 160 of them with total cholesterol> 200 mg/dl participated in the study. They were randomized with a 2:1 ratio of receiving CMO capsules (containing 200 mg mastiha oil per capsule) and placebo for a total of 8 weeks respectively. 113 patients received CMO and 47 were randomized in the control group, and all of them completed the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

- Increased total cholesterol >200 mg/dl, in adult volunteers (≥18 years old) of any gender, not amenable or not willing to receive pharmaceutical therapy.

Exclusion Criteria:

* Participation in any other study during the recruitment period
* Contribution in the design or accomplishment of the study
* Known cardiovascular disease (coronary artery disease, carotid artery disease, peripheral vascular disease, stroke, diabetes mellitus, aortic aneurysm)
* Patients in high or very high risk of CVD according to SCORE2
* Subjects amenable to pharmaceutical lipid-lowering regimens according to current guideline, or any other pharmaceutical regimen with hypolipidemic effects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Total cholesterol | 8 weeks
  Decrease in total cholesterol serum levels
LDL cholesterol | 8 weeks
  Decrease in LDL cholesterol serum levels
HDL cholesterol | 8 weeks
  Increase in HDL cholesterol serum levels
Triglycerides | 8 weeks
  Decrease in triglycerides serum levels

SECONDARY OUTCOMES:
Glucose | 8 weeks
  Decrease in glucose serum levels
Liver tests | 8 weeks
  Change in liver tests (SGOT, SGPT, gGT)
Renal tests | 8 weeks
  Change in renal tests (BUN, creatinine)
Electrolytes | 8 weeks
  Change in electrolyte levels (sodium, potassium)
Inflammation markers | 8 weeks
  Change in inflammation markers tests (CRP, uric acid)

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Kartalis, MD, Principal Investigator — Skylitseio General Hospital of Chios, Greece; Matthaios Didagelos, MD, PhD, Principal Investigator — AHEPA University General Hospital, Thessaloniki, Greece
Locations (1):
- Skylitseio General Hospital, Chios, Greece

IPD SHARING:
Plan to Share IPD: No